CLINICAL TRIAL: NCT02408926
Title: Vaccine Responses in Infants After Acellular Pertussis Vaccination During Pregnancy in Thailand
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Chulalongkorn University (Other); Institut Pasteur de Lille (Other); Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Elke Leuridan, MD, PhD, Prof., MD, PhD, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: cev002
Record Dates: First submitted 2015-03-23; First posted 2015-04-06 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Pertussis
Keywords: Pertussis; Pregnancy; Humoral immune response; Functionality; Vaccination
MeSH Terms: conditions — Whooping Cough | interventions — Boostrix; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Poliovirus Vaccine, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Women will be vaccinated with an acellular pertussis containing vaccine (Boostrix) between 27 and 36 weeks of gestation. Children born from these mothers will be vaccinated according to the official recommendations in Thailand at 2, 4, 6 and 18 months with a hexavalent acellular pertussis containing vaccine (Infanrix hexa).
  Interventions: Biological: Boostrix; Biological: Infanrix hexa
- Group B (Active Comparator): Women will be vaccinated with an acellular pertussis containing vaccine (Boostrix) between 27 and 36 weeks of gestation. Children born from these mothers will be vaccinated according to the official recommendations in Thailand at 2, 4, 6 and 18 months with a pentavalent whole cell pertussis containing vaccine (Quinvaxem). OPV (oral poliovirus vaccine) will also be administered at 2, 4, 6 and 18 months.
  Interventions: Biological: Boostrix; Biological: Quinvaxem; Biological: OPV

INTERVENTIONS:
Biological: Boostrix — Pregnant women will be vaccinated with an acellular pertussis containing vaccine between 27 and 36 weeks of gestation.
  Other Names: Acellular pertussis containing vaccine
Biological: Infanrix hexa — Children from group A will be vaccinated with an acellular pertussis containing vaccine according to the official recommendations in Thailand at 2, 4, 6 and 18 months.
  Other Names: Acellular pertussis containing vaccine
  Arms: Group A
Biological: Quinvaxem — Children from group B will be vaccinated with a whole cell pertussis containing vaccine according to the official recommendations in Thailand at 2, 4, 6 and 18 months.
  Other Names: Whole cell pertussis containing vaccine
  Arms: Group B
Biological: OPV — Children from group B will be vaccinated with OPV vaccine according to the official recommendations in Thailand at 2, 4, 6 and 18 months.
  Other Names: Oral Polio Vaccine
  Arms: Group B

SUMMARY:
Young infants are most vulnerable to severe disease and even death when infected with Bordetella pertussis. The current vaccines and vaccination programs do not guarantee protection of neonates from this disease. Maternal acquired pertussis-specific antibodies show low concentrations with short persistence in newborns creating a susceptibility gap for infection between birth and the first vaccinations. A possible strategy to protect infants from birth is pertussis vaccination during pregnancy, which will increase the amount of passively transferred maternal antibodies.

However, little is known regarding the effect of high titers of maternal antibodies on the infants immune responses to different pertussis vaccines (whole cell versus acellular). Humoral immune responses will be assessed in infants receiving whole cell versus infants receiving acellular pertussis vaccines. Functionality of the antibodies will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Willing to be immunized with a pertussis containing vaccine during pregnancy
* Intend to be available for follow-up visits and phone call through 19 months postpartum
* Willing to have infant immunized with a pertussis containing vaccine at 2, 4, 6 months and 18 months of age according to EPI (Expanded Programme of Immunization) and receiving (randomized) either acellular pertussis (aP) (study vaccine) or a whole cell pertussis (wP) vaccine. Consent for participation of the child is needed by both married parents or by a single unmarried other.
* At low risk for pregnancy related complications as determined by the investigator and a second trimester ultrasound with no significant abnormalities.

Exclusion Criteria:

Pregnant subjects

* Multiple pregnancies
* Serious obstetrical risk
* Serious underlying medical condition
* Significant mental illness
* History of febrile illness (greater than or equal to 38°C) within the past 72 hours before injection
* Previous severe reaction to any vaccine
* Receipt of tetanus-diphtheria toxoid immunization within the past 1 month Receipt of an pertussis containing vaccine (Tdap) in the last 5 years
* Receipt of a vaccine, blood product (excluding Rhogam) within the 4 weeks prior to injection through 4 weeks following injection and IVIG (Intravenous Immunoglobulins) within 12 weeks period. One month interval should be respected with another vaccine (except influenza) in orde to evaluate Adverse events following one or both vaccines (fever, local symptoms)
* Receipt of an experimental drug during pregnancy
* Anything in the opinion of the investigator that would prevent women from completing the study or put the woman at risk

Infants

* Preterm delivery before 37 weeks of gestation
* Serious underlying medical condition
* Children suffering from primary humoral immune disorders; suffering from primary cellular immune deficiencies and disorders from the complete cascade
* No informed consent from one or both married parents
* Severe reactions to any vaccine
* Anything in the opinion of the investigator that would prevent children from completing the study or put the child at risk

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 370 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
kinetics of Pertussis toxin (PT) IgG titers in infants | from birth until 19 months of age
  Measurement of anti- Pertussis Toxin (PT) immunoglobulin (IgG) antibodies at several time points following maternal vaccination during pregnancy and after infant immunization (priming and boosting) with an acellular or whole cell pertussis containing vaccine
kinetics of Filamentous haemagglutinin (FHA) IgG titers in infants | from birth until 19 months of age
  Measurement of anti- Filamentous Haemmaglutinin (FHA) immunoglobulin (IgG) antibodies at several time points following maternal vaccination during pregnancy and after infant immunization (priming and boosting) with an acellular or whole cell pertussis containing vaccine
kinetics of Pertactin (Prn) IgG titers in infants | from birth until 19 months of age
  Measurement of anti- Pertactin (Prn) immunoglobulin (IgG) antibodies at several time points following maternal vaccination during pregnancy and after infant immunization (priming and boosting) with an acellular or whole cell pertussis containing vaccine

SECONDARY OUTCOMES:
Functionality of the maternal anti-PT IgG antibodies in the infants as assessed with a newly validated luminescence based assay | At birth
  functionality of the passively acquired anti-PT antibodies in infants following maternal vaccination during pregnancy with an acellular pertussis containing vaccine (Boostrix), as assessed with a newly validated luminescence based assay
Functionality of the anti-PT IgG antibodies in the infants after vaccination assessed with a newly validated luminescence based assay | At month 7 and month 19
  To measure the functionality of the anti-PT antibodies in infants vaccinated with either an acellular pertussis containing vaccine (Infanrix hexa) or a whole cell pertussis vaccine (Quinvaxem), after maternal vacicnation during pregnancy, assessed with a newly validated luminescence based assay
Efficacy of the transplacental transport of IgG as assessed by the ratio of cord and maternal titers of IgG antibodies | Birth
  Efficacy as assessed by the ratio of cord and maternal titers of IgG antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Elke Leuridan, MD PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

REFERENCES:
- [Derived] Wanlapakorn N, Sarawanangkoor N, Srimuan D, Thatsanathorn T, Klinfueng S, Poovorawan Y. Persistence of hepatitis B surface antibody until 7 years of age following administration of hexavalent and pentavalent vaccines in children at 2, 4, 6, and 18 months. Vaccine X. 2024 Sep 20;20:100561. doi: 10.1016/j.jvacx.2024.100561. eCollection 2024 Oct. PMID 39385752
- [Derived] Sarawanangkoor N, Wanlapakorn N, Srimuan D, Thatsanathorn T, Thongmee T, Poovorawan Y. Persistence of Antibodies against Measles, Mumps, and Rubella after the Two-Dose MMR Vaccination: A 7-Year Follow-Up Study. Vaccines (Basel). 2024 Jul 5;12(7):744. doi: 10.3390/vaccines12070744. PMID 39066382
- [Derived] Wanlapakorn N, Sarawanangkoor N, Srimuan D, Thatsanathorn T, Thongmee T, Poovorawan Y. Antibody persistence to diphtheria toxoid, tetanus toxoid, Bordetella pertussis antigens, and Haemophilus influenzae type b following primary and first booster with pentavalent versus hexavalent vaccines. Hum Vaccin Immunother. 2024 Dec 31;20(1):2352909. doi: 10.1080/21645515.2024.2352909. Epub 2024 May 16. PMID 38752802
- [Derived] Embacher S, Maertens K, Herzog SA. Half-life Estimation of Pertussis-Specific Maternal Antibodies in (Pre)Term Infants After In-Pregnancy Tetanus, Diphtheria, Acellular Pertussis Vaccination. J Infect Dis. 2023 Nov 28;228(11):1640-1648. doi: 10.1093/infdis/jiad212. PMID 37285482
- [Derived] Hu S, Logan N, Puenpa J, Wanlapakorn N, Vongpunsawad S, Poovorawan Y, Willett BJ, Hosie MJ. Evaluation of the effect of maternally derived antibody on response to MMR vaccine in Thai infants. Vaccine. 2022 Mar 1;40(10):1439-1447. doi: 10.1016/j.vaccine.2022.01.049. Epub 2022 Feb 5. PMID 35135700
- [Derived] Wanlapakorn N, Puenpa J, Thongmee T, Srimuan D, Thatsanathorn T, Vongpunsawad S, Poovorawan Y. Antibodies to measles, mumps, and rubella virus in Thai children after two-dose vaccination at 9 months and 2.5 years: A longitudinal study. Vaccine. 2020 May 19;38(24):4016-4023. doi: 10.1016/j.vaccine.2020.04.013. Epub 2020 Apr 21. PMID 32331806
- [Derived] Wanlapakorn N, Maertens K, Vongpunsawad S, Puenpa J, Tran TMP, Hens N, Van Damme P, Thiriard A, Raze D, Locht C, Poovorawan Y, Leuridan E. Quantity and Quality of Antibodies After Acellular Versus Whole-cell Pertussis Vaccines in Infants Born to Mothers Who Received Tetanus, Diphtheria, and Acellular Pertussis Vaccine During Pregnancy: A Randomized Trial. Clin Infect Dis. 2020 Jun 24;71(1):72-80. doi: 10.1093/cid/ciz778. PMID 31418814